CLINICAL TRIAL: NCT06031233
Title: Evaluating the Safety of Shortened Infusion Times for dIfferent Oncological Immunotherapies; An Observational Prospective Study
Brief Title: Evaluating the Safety of Shortened Infusion Times for dIfferent Oncological Immunotherapie
Acronym: MINUTE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, HB Fiebrich-Westra, Principal Investigator, Isala
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83071.075.22 / 20221102
Record Dates: First submitted 2023-04-24; First posted 2023-09-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-10

CONDITIONS: Oncology; Infusion Reaction
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; pembrolizumab; Ipilimumab; durvalumab; atezolizumab; Bevacizumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Nivolumab (Experimental): If no infusion reaction has occurred after 2 cyclues, infusion time will stepwise be shortened to 10 minutes in the following cycles.
  Interventions: Drug: Nivolumab
- Pembrolizumab (Experimental): If no infusion reaction has occurred after 2 cyclues, infusion time will stepwise be shortened to 10 minutes in the following cycles.
  Interventions: Drug: Pembrolizumab
- ipilimumab (Experimental): If no infusion reaction has occurred after 2 cyclues, infusion time will stepwise be shortened to 10 minutes in the following cycles.
  Interventions: Drug: Ipilimumab
- Durvalumab (Experimental): If no infusion reaction has occurred after 2 cyclues, infusion time will stepwise be shortened to 10 minutes in the following cycles.
  Interventions: Drug: Durvalumab
- Atezolizumab (Experimental): If no infusion reaction has occurred after 2 cyclues, infusion time will stepwise be shortened to 10 minutes in the following cycles.
  Interventions: Drug: Atezolizumab
- bevacizumab (Experimental): If no infusion reaction has occurred after 2 cyclues, infusion time will stepwise be shortened to 10 minutes in the following cycles.
  Interventions: Drug: Bevacizumab
- Trastuzumab (Experimental): If no infusion reaction has occurred after 2 cyclues, infusion time will stepwise be shortened to 10 minutes in the following cycles.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Nivolumab — Gradual shortening of infusion times
  Arms: Nivolumab
Drug: Pembrolizumab — Gradual shortening of infusion times
  Arms: Pembrolizumab
Drug: Ipilimumab — Gradual shortening of infusion times
  Arms: ipilimumab
Drug: Durvalumab — Gradual shortening of infusion times
  Arms: Durvalumab
Drug: Atezolizumab — Gradual shortening of infusion times
  Arms: Atezolizumab
Drug: Bevacizumab — Gradual shortening of infusion times
  Arms: bevacizumab
Drug: Trastuzumab — Gradual shortening of infusion times
  Arms: Trastuzumab

SUMMARY:
This study is an interventional, explorative, prospective study to show whether shortening of infusion times for patients using nivolumab, pembrolizumab, ipilimumab, trastuzumab, bevacizumab, durvalumab or atezolizumab continues to be associated with an acceptable safety profile.

Infusion times will be gradually shortened if tolerability allowes.

DETAILED DESCRIPTION:
After two cycles with normal infusion times, infusion time will be shortened to 15 mintues en 10 minutes subsequently if no infusion reaction occurs.

Patient satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Starting treatment with monoclonal antibodies: nivolumab, pembrolizumab ipilimumab, bevacizumab, trastuzumab, durvalumab or atezolizumab.
* 18 years and older.
* No known history of increased susceptibility to immunological reactions.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.

Exclusion Criteria:

* Other research medication within 4 weeks of the start of the study.
* Inclusion in medical research in which the administration of medication should follow its stated times and dosages of infusions
* Dosage deviates from standard protocol
* Patients whom receive drugs through a central venous catheter (and for example porth-a-cath).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of infusion related reactions | During or within 30 minutes after the end of the infusion

SECONDARY OUTCOMES:
Plasma levels of the administered mAb | Within 15 minutes before start of the infusion

OTHER OUTCOMES:
Satisfaction with shortened infusion time assessed by the VAS | Directly after infusion in fourth cycle (cycle length ranges from 21-42 days, depending on the specific antibody)
  Scale 1-10, 1: not satisfied at all, 10: most satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Isala Hospital, Zwolle, Netherlands

IPD SHARING:
Plan to Share IPD: No